CLINICAL TRIAL: NCT05218499
Title: Brightline-1: A Phase II/III, Randomized, Open-label, Multi-center Study of Brigimadlin (BI 907828) Compared to Doxorubicin as First Line Treatment of Patients With Advanced Dedifferentiated Liposarcoma
Brief Title: Brightline-1: A Study to Compare Brigimadlin (BI 907828) With Doxorubicin in People With a Type of Cancer Called Dedifferentiated Liposarcoma
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1403-0008; 2021-002392-20 (EudraCT Number)
Record Dates: First submitted 2022-01-18; First posted 2022-02-01 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Liposarcoma, Dedifferentiated
MeSH Terms: conditions — Liposarcoma | interventions — brigimadlin; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Brigimadlin 30 mg q3w (Experimental): Patients with advanced or metastatic dedifferentiated liposarcoma (DDLPS) received 30 milligram (mg) brigimadlin taken orally on day 1 of each 21-day cycle (q3w).
  Interventions: Drug: Brigimadlin
- Brigimadlin 45 mg q3w (Experimental): Patients with advanced or metastatic dedifferentiated liposarcoma (DDLPS) received 45 milligram (mg) brigimadlin taken orally on day 1 of each 21-day cycle (q3w).
  Interventions: Drug: Brigimadlin
- Doxorubicin (Active Comparator): Patients with advanced or metastatic dedifferentiated liposarcoma (DDLPS) received one intravenous infusion of 75 milligram per square meter (mg/m2) on Day 1 of each 21-day cycle (q3w) until a maximum cumulative dose of 450 mg/m2 (approximately 6 cycles).
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Brigimadlin — Brigimadlin taken orally on day 1 of each 21-day cycle (q3w).
  Other Names: BI 907828
  Arms: Brigimadlin 30 mg q3w; Brigimadlin 45 mg q3w
Drug: Doxorubicin — Intravenous infusion of 75 milligram per square meter (mg/m2) on Day 1 of each 21-day cycle (q3w) until a maximum cumulative dose of 450 mg/m2 (approximately 6 cycles).
  Arms: Doxorubicin

SUMMARY:
This study is open to people with a type of cancer called dedifferentiated liposarcoma. People with advanced liposarcoma aged 18 or older who are not receiving any other cancer treatment can participate.

The purpose of this study is to compare a medicine called brigimadlin (BI 907828) with doxorubicin in people with liposarcoma. Brigimadlin (BI 907828) is a so-called MDM2 inhibitor that is being developed to treat cancer. Doxorubicin is a medicine already used to treat cancer including liposarcoma.

During the study, participants get either brigimadlin (BI 907828) or doxorubicin. Every 3 weeks, participants take brigimadlin (BI 907828) as tablets or doxorubicin as an infusion into a vein. Participants can switch to brigimadlin (BI 907828) treatment if they did not benefit from doxorubicin treatment.

Participants can continue treatment in the study as long as they benefit from it and can tolerate it.

Doctors regularly check the size of the tumour and check whether it has spread to other parts of the body. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated, written informed consent form (ICF) in accordance with ICH-GCP and local legislation prior to any trial-specific procedures, sampling, or analyses.
* Male or female patients ≥18 years old at the time of signature of the informed consent form (ICF). Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use 2 medically acceptable methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly beginning at screening, during trial participation, and until 6 months and 12 days after last dose for women and 102 days after last dose for men. A list of contraception methods meeting these criteria is provided in the patient information.
* Histologically proven locally advanced or metastatic, unresectable (surgery morbidity would outweigh potential benefits), progressive or recurrent dedifferentiated liposarcoma (DDLPS). Locally performed histopathological diagnosis will be accepted for entry into this trial but will be confirmed by independent pathological review while the patients receive treatment in this trial.
* Written pathology report indicating the diagnosis of DDLPS with positive mouse double minute 2 homolog (MDM2) immunohistochemistry or MDM2 amplification as demonstrated by fluorescence in situ hybridization or next generation sequencing (NGS) must be available.
* Formalin fixed paraffin embedded tumor blocks or slides must be available for retrospective histopathological central review.
* Presence of at least one measurable target lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. In patients who only have one target lesion, the baseline imaging must be performed at least 2 weeks after any biopsy of the target lesion.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Patient must be willing to donate blood samples for the pharmacokinetics, pharmacodynamics, and tumor mutation analysis.
* Patient willing to undergo a mandatory tumor biopsy at the time point specified in the flowchart unless exempt.
* Adequate organ function.

Exclusion Criteria:

* Known mutation in the TP53 gene (screening for TP53 status is not required).
* Major surgery (major according to the investigator's assessment) performed within 4 weeks prior to randomization or planned within 6 months after screening.
* Prior systemic therapy for liposarcoma in any setting (including adjuvant, neoadjuvant, maintenance, palliative).
* Previous or concomitant malignancies other than DDLPS or WDLPS, treated within the previous 5 years, except effectively treated non-melanoma skin cancers, carcinoma in situ of the cervix, ductal carcinoma in situ, or other malignancy that is considered cured by local treatment.
* Previous treatment with anthracyclines in any setting (systemic treatment with other anticancer agents is allowed if completed at least 5 years prior to study entry with the exception of hormone therapy).
* Patients who must or intend to continue the intake of restricted medications or any drug considered likely to interfere with the safe conduct of the trial.
* Currently enrolled in another investigational device or drug trial, or less than 30 days since ending another investigational device or drug trial(s) or receiving other investigational treatment(s).
* Patients not expected to comply with the protocol requirements or not expected to complete the trial as scheduled (e.g. chronic alcohol or drug abuse or any other condition that, in the investigator's opinion, makes the patient an unreliable trial participant).
* Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2026-01-29 (Estimated)

CONTACTS AND LOCATIONS:
Locations (109):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - Precision NextGen Oncology, Beverly Hills, California
  - City of Hope-Duarte-56419, Duarte, California
  - University of Southern California, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Mayo Clinic Cancer Center, Jacksonville, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Nebraska Cancer Specialists-Omaha-69502, Omaha, Nebraska
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Prince of Wales Hospital-Randwick-66496, Randwick, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- UZ Leuven, Leuven, Belgium
- Canada (4):
  - BC Cancer Agency - Vancouver, Vancouver, British Columbia
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- China (9):
  - Cancer Hospital of Chinese Academy of Medical Science, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - West China Hospital of Sichuan University, Chengdu
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongshan Hospital Affiliated to Fudan University, Shanghai
  - Wuhan Union Hospital, Wuhan
- Czechia (3):
  - Masaryk Memorial Cancer Institute, Brno
  - University Hospital Olomouc, Olomouc
  - University Hospital Motol, Prague
- Herlev and Gentofte Hospital, Herlev, Denmark
- Finland (2):
  - HUCH Comprehensive Cancer Center, building 2, Helsinki
  - Tampere University Hospital, Tampere
- France (8):
  - INS Bergonie, Bordeaux
  - CTR Oscar Lambret, Lille
  - CTR Leon Berard, Lyon
  - HOP Timone, Marseille
  - Hôpital Cochin, Paris
  - CTR Eugène Marquis, Rennes
  - INS Claudius Regaud IUCT-Oncopole, Toulouse
  - INS Gustave Roussy, Villejuif
- Germany (9):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Helios Klinikum Berlin-Buch, Berlin
  - Technische Universität Dresden, Dresden
  - Universitätsklinikum Essen AöR, Essen
  - Asklepios Kliniken GmbH & Co. KGaA, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Klinikum der Universität München AÖR, München
  - Robert Bosch Gesellschaft für medizinische Forschung mbH, Stuttgart
- Greece (3):
  - Hippokration General Hospital of Athen, Athens
  - "Attikon" University General Hospital of Attica, Haidari
  - Bioclinic Thessaloniki, Thessaloniki
- Prince of Wales Hospital-Hong Kong-20715, Hong Kong, Hong Kong
- Italy (8):
  - Humanitas Gavazzeni, Bergamo
  - Istituto Di Candiolo, Candiolo (TO)
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli
  - AOU San Luigi Gonzaga, Orbassano (TO)
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Università Campus Bio-Medico - ROMA, Roma
- Japan (11):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - Nagoya University Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Tohoku University Hospital, Miyagi, Sendai
  - Okayama University Hospital, Okayama, Okayama
  - Osaka International Cancer Institute, Osaka, Osaka
  - Hokkaido Cancer Center, Sapporo, Hokkaido
  - National Cancer Center Hospital, Tokyo, Chuo-ku
  - Japanese Foundation for Cancer Research, Tokyo, Koto-ku
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Leids Universitair Medisch Centrum (LUMC), Leiden
- Oslo Universitetssykehus HF, Radiumhospitalet, Oslo, Norway
- Portugal (2):
  - IPO Lisboa Francisco Gentil, EPE, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
- Spain (10):
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital Miguel Servet, Zaragoza
- Sweden (2):
  - Skånes universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset Stockholm, Stockholm
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)
- United Kingdom (5):
  - Addenbrooke's Hospital, Cambridge
  - Velindre Cancer Centre, Cardiff
  - Churchill Hospital, Headington
  - University College Hospital, London
  - The Royal Marsden Hospital, Chelsea, London

IPD SHARING:
Plan to Share IPD: Yes
Once the time frame criteria given under number 4 are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Schoffski P, Lahmar M, Lucarelli A, Maki RG. Brightline-1: phase II/III trial of the MDM2-p53 antagonist BI 907828 versus doxorubicin in patients with advanced DDLPS. Future Oncol. 2023 Mar;19(9):621-629. doi: 10.2217/fon-2022-1291. Epub 2023 Mar 29. PMID 36987836
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, active-controlled, open-label, global trial with a seamless Phase II part and Phase III part parallel design.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin
Started | 90 | 148 | 162
Doxorubicin Patients Who Crossed Over to Brigimadlin 30 mg q3w | 0 | 0 | 7 (Patients who had a confirmed Progressive Disease after receiving doxorubicin and then cross-over to treatment with brigimadlin 30 mg q3w.)
Doxorubicin Patients Who Crossed Over to Brigimadlin 45 mg q3w | 0 | 0 | 70 (Patients who had a confirmed Progressive Disease after receiving doxorubicin and then cross-over to treatment with brigimadlin 45 mg q3w.)
Completed | 0 | 0 | 76 (Completed planned treatment period)
Not Completed | 90 | 148 | 86
Not completed — Not treated | 1 | 1 | 8
Not completed — Death | 2 | 0 | 0
Not completed — Other than listed | 3 | 7 | 10
Not completed — Protocol deviation | 5 | 6 | 4
Not completed — Technical problems | 0 | 1 | 0
Not completed — Burden of trial procedures | 0 | 1 | 2
Not completed — Clinical disease progression | 6 | 6 | 11
Not completed — Objective disease progression | 44 | 61 | 42
Not completed — Adverse Event | 11 | 36 | 9
Not completed — On treatment at time of snapshot | 18 | 29 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized, regardless of whether they have received any trial medication or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin | Total
Number analyzed (Participants) | 90 | 148 | 162 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (11.7) | 64.7 (9.8) | 63.0 (11.7) | 63.5 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 52 | 62 | 149
  Male | 55 | 96 | 100 | 251
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 9 | 23
  Not Hispanic or Latino | 79 | 138 | 150 | 367
  Unknown or Not Reported | 3 | 4 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 20 | 39 | 29 | 88
  Black or African American | 1 | 1 | 2 | 4
  White | 65 | 103 | 128 | 296
  Missing | 3 | 5 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) based on blinded central independent review. For each patient, PFS was defined as the time interval from randomization until tumor progression according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (solely based on blinded central independent review) or death from any cause, whichever occurs first.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 20.6 months.
Population: Randomised Set (RS): All patients randomized, regardless of whether they have received any trial medication or not.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin
Number analyzed (Participants) | 90 | 148 | 162
Months | 8.18 [2.96 to 16.66] | 8.38 [3.94 to NA] — Not evaluable: not enough events reached. | 7.16 [2.63 to 11.33]
Statistical Analysis 1: Comparison: Brigimadlin 30 mg q3w vs Brigimadlin 45 mg q3w vs Doxorubicin; The primary estimator for the hazard ratio is the median unbiased estimator. The confidence interval (CI) for the hazard ratio is calculated as a repeated CI. The p-value is obtained using a weighted inverse normal method combining one-sided p-values from two stages; Test type: Other; p = 0.0956, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.60 to 1.06] — A hazard ratio value below 1 favors brigimadlin

2. Secondary Outcome: Objective Response (OR)
Description: Objective response (OR), defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.1 (based on blinded central independent review) from the date of randomization until disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent, whichever occurs first.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 20.6 months.
Population: Randomised Set (RS): All patients randomized, regardless of whether they have received any trial medication or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin
Number analyzed (Participants) | 90 | 148 | 162
Participants | 13 | 33 | 14
Statistical Analysis 1: Comparison: Brigimadlin 30 mg q3w vs Brigimadlin 45 mg q3w vs Doxorubicin; The primary estimator and CI for the odds ratio is by Cochran-Mantel-Haenszel; Test type: Other; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.52 to 5.67] — An odds ratio value greater than 1 favors brigimadlin

3. Secondary Outcome: Duration of Objective Response (DOR)
Description: Duration of objective response (DOR), defined as the time interval from first documented confirmed OR until disease progression or death among patients with confirmed OR (based on blinded central independent review), whichever occurs first.
Time Frame: Up to 20.6 months.
Population: All patients randomized who had an objective response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin
Number analyzed (Participants) | 13 | 33 | 14
Months | NA [8.51 to NA] — Not enough participants with events. | 9.92 [9.72 to NA] — Not enough participants with events. | 9.99 [9.89 to 15.41]

4. Secondary Outcome: Disease Control (DC)
Description: Disease control (DC), defined as a best overall response of CR, PR, or stable disease (SD) according to RECIST version 1.1 (based on blinded central independent review).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Up to 20.6 months.
Population: Randomised Set (RS): All patients randomized, regardless of whether they have received any trial medication or not.
Measure: Count of Participants; unit: Participants
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin
Number analyzed (Participants) | 90 | 148 | 162
Participants | 71 | 128 | 117
Statistical Analysis 1: Comparison: Brigimadlin 30 mg q3w vs Doxorubicin; Odds ratios are calculated from a logistic regression model with the stratification factor (locally advanced vs. metastatic) included as a covariate; Test type: Other; Odds Ratio (OR) = 1.51, 95% CI 2-sided [0.81 to 2.82] — An odds ratio value greater than 1 favors brigimadlin
Statistical Analysis 2: Comparison: Brigimadlin 45 mg q3w vs Doxorubicin; Odds ratios are calculated from a logistic regression model with the stratification factor (locally advanced vs. metastatic) included as a covariate. Exact 95% confidence interval (CI) by Clopper and Pearson; Test type: Other; Odds Ratio (OR) = 2.67, 95% CI 2-sided [1.48 to 4.84] — An odds ratio value greater than 1 favors brigimadlin

5. Secondary Outcome: Change in Health-Related Quality of Life at Week 6 and 18
Description: Mean change from baseline to week 6 and 18 in the following European Organization for Research and Treatment on Cancer (EORTC) Quality of Life Core Questionnaire 30 items (QLQ-C30) scores:
  * Physical functioning (higher score is better)
  * Pain (higher score is worse)
  * Fatigue (higher score is worse)
  * Global health status / QoL (higher score is better)
  and the following scores obtained using items from the EORTC QLQ-C30 and EORTC Item Library (higher score is worse):
  * Fatigue symptoms
  * Fatigability
  * Fatigue impact
  * Pain descriptors
  * Pain impact
  All of the scales and single-item measures range in score from 0 to 100.
Time Frame: Baseline (cycle 1 day 1), week 6 and week 18.
Population: Randomised Set (RS). As per protocol, the endpoint was performed as part of the Phase III of the trial, which only includes the selected investigational arm (brigimadlin 45 mg q3w) and the doxorubicin control arm.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Brigimadlin 45 mg q3w | Doxorubicin
Number analyzed (Participants) | 121 | 114
Score on a scale
  Physical functioning - Change from baseline at Week 6: number analyzed (Participants) | 94 | 85
  Physical functioning - Change from baseline at Week 6 | -2.1 (17.4) | -5.5 (17.9)
  Physical functioning - Change from baseline at Week 18: number analyzed (Participants) | 69 | 49
  Physical functioning - Change from baseline at Week 18 | -5.9 (20.8) | -7.5 (16.3)
  Pain - Change from baseline at Week 6: number analyzed (Participants) | 94 | 85
  Pain - Change from baseline at Week 6 | -3.7 (20.2) | 0.8 (25.2)
  Pain - Change from baseline at Week 18: number analyzed (Participants) | 69 | 49
  Pain - Change from baseline at Week 18 | 1.4 (26.0) | -1.0 (26.7)
  Fatigue - Change from baseline at Week 6: number analyzed (Participants) | 94 | 85
  Fatigue - Change from baseline at Week 6 | 3.4 (21.2) | 10.5 (23.5)
  Fatigue - Change from baseline at Week 18: number analyzed (Participants) | 69 | 49
  Fatigue - Change from baseline at Week 18 | 8.1 (27.5) | 14.1 (27.5)
  Global health status / quality of life - Change from baseline at Week 6: number analyzed (Participants) | 94 | 85
  Global health status / quality of life - Change from baseline at Week 6 | -0.6 (18.6) | -8.9 (22.4)
  Global health status / quality of life - Change from baseline at Week 18: number analyzed (Participants) | 69 | 49
  Global health status / quality of life - Change from baseline at Week 18 | -5.8 (24.5) | -8.0 (20.8)
  Fatigue symptoms - Change from baseline at Week 6: number analyzed (Participants) | 100 | 90
  Fatigue symptoms - Change from baseline at Week 6 | 3.4 (19.2) | 10.6 (25.1)
  Fatigue symptoms - Change from baseline at Week 18: number analyzed (Participants) | 75 | 52
  Fatigue symptoms - Change from baseline at Week 18 | 7.9 (26.7) | 14.7 (26.2)
  Fatigability - Change from baseline at Week 6: number analyzed (Participants) | 100 | 90
  Fatigability - Change from baseline at Week 6 | 3.3 (19.8) | 11.2 (21.8)
  Fatigability - Change from baseline at Week 18: number analyzed (Participants) | 75 | 52
  Fatigability - Change from baseline at Week 18 | 5.1 (23.3) | 16.4 (24.3)
  Fatigue impact - Change from baseline at Week 6: number analyzed (Participants) | 100 | 90
  Fatigue impact - Change from baseline at Week 6 | -1.5 (20.5) | 3.5 (23.7)
  Fatigue impact - Change from baseline at Week 18: number analyzed (Participants) | 75 | 52
  Fatigue impact - Change from baseline at Week 18 | 1.6 (23.5) | 6.2 (25.9)
  Pain descriptors - Change from baseline at Week 6: number analyzed (Participants) | 96 | 85
  Pain descriptors - Change from baseline at Week 6 | -2.7 (18.5) | 0.9 (16.5)
  Pain descriptors - Change from baseline at Week 18: number analyzed (Participants) | 71 | 50
  Pain descriptors - Change from baseline at Week 18 | 0.4 (24.1) | 1.8 (17.7)
  Pain impact - Change from baseline at Week 6: number analyzed (Participants) | 96 | 85
  Pain impact - Change from baseline at Week 6 | -3.0 (14.7) | 1.9 (18.9)
  Pain impact - Change from baseline at Week 18: number analyzed (Participants) | 71 | 50
  Pain impact - Change from baseline at Week 18 | 0.6 (19.6) | 2.4 (20.5)

ADVERSE EVENTS:
Time Frame: Up to approximately 20.8 months.
Description: This patient set includes all patients who were documented to have taken at least one dose of trial medication (brigimadlin or doxorubicin).
Groups:
- Doxorubicin - Brigimadlin 30 mg q3w: Patients on Doxorubicin with a confirmed disease progression who crossed to Brigimadlin 30 mg taken orally on day 1 of each 21-day cycle (q3w).
- Doxorubicin - Brigimadlin 45 mg q3w: Patients on Doxorubicin with a confirmed disease progression who crossed to Brigimadlin 45 mg taken orally on day 1 of each 21-day cycle (q3w).
Arm/Group | Brigimadlin 30 mg q3w | Brigimadlin 45 mg q3w | Doxorubicin | Doxorubicin - Brigimadlin 30 mg q3w | Doxorubicin - Brigimadlin 45 mg q3w
All-Cause Mortality (participants affected / at risk) | 31/89 | 40/147 | 15/154 | 5/7 | 22/70
Serious Adverse Events (participants affected / at risk) | 27/89 | 57/147 | 42/154 | 1/7 | 22/70
Other Adverse Events (participants affected / at risk) | 89/89 | 144/147 | 153/154 | 6/7 | 67/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brigimadlin 30 mg q3w (N=89) | Brigimadlin 45 mg q3w (N=147) | Doxorubicin (N=154) | Doxorubicin - Brigimadlin 30 mg q3w (N=7) | Doxorubicin - Brigimadlin 45 mg q3w (N=70)
Anaemia (Blood and lymphatic system disorders) | 1 | 7 | 2 | 0 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 12 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 6 | 2 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Duodenal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 0 | 0 | 1
Disease progression (General disorders) | 1 | 0 | 1 | 0 | 2
Fatigue (General disorders) | 0 | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 0
Hyperthermia (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 2 | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 4 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Focal peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Fungaemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Phlebitis infective (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 3 | 2 | 0 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 5 | 4 | 0 | 0
Platelet count decreased (Investigations) | 1 | 12 | 2 | 0 | 1
Troponin I increased (Investigations) | 0 | 0 | 1 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 2 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0 | 0 | 0
Device physical property issue (Product Issues) | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Obstructive nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 0
Renal vein embolism (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Ovarian vein thrombosis (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 7 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Assisted suicide (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Aortic thrombosis (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3 | 2 | 0 | 2
Embolism (Vascular disorders) | 0 | 4 | 1 | 0 | 1
Embolism arterial (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Pelvic venous thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Superficial vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brigimadlin 30 mg q3w (N=89) | Brigimadlin 45 mg q3w (N=147) | Doxorubicin (N=154) | Doxorubicin - Brigimadlin 30 mg q3w (N=7) | Doxorubicin - Brigimadlin 45 mg q3w (N=70)
Anaemia (Blood and lymphatic system disorders) | 22 | 52 | 63 | 1 | 22
Leukopenia (Blood and lymphatic system disorders) | 2 | 15 | 21 | 0 | 3
Lymphopenia (Blood and lymphatic system disorders) | 2 | 4 | 6 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 16 | 42 | 49 | 1 | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 40 | 10 | 0 | 15
Palpitations (Cardiac disorders) | 1 | 4 | 2 | 0 | 4
Hypoacusis (Ear and labyrinth disorders) | 1 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 5 | 7 | 3 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 18 | 28 | 18 | 0 | 14
Abdominal pain upper (Gastrointestinal disorders) | 10 | 7 | 9 | 0 | 2
Constipation (Gastrointestinal disorders) | 20 | 26 | 37 | 0 | 11
Diarrhoea (Gastrointestinal disorders) | 35 | 60 | 42 | 2 | 24
Dry mouth (Gastrointestinal disorders) | 3 | 8 | 3 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 12 | 8 | 11 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 8 | 6 | 0 | 1
Nausea (Gastrointestinal disorders) | 71 | 112 | 90 | 4 | 46
Stomatitis (Gastrointestinal disorders) | 2 | 7 | 33 | 0 | 4
Vomiting (Gastrointestinal disorders) | 47 | 55 | 28 | 2 | 21
Asthenia (General disorders) | 29 | 32 | 40 | 1 | 18
Fatigue (General disorders) | 30 | 65 | 56 | 3 | 18
Influenza like illness (General disorders) | 2 | 5 | 2 | 1 | 4
Malaise (General disorders) | 7 | 14 | 12 | 0 | 5
Mucosal inflammation (General disorders) | 2 | 7 | 22 | 0 | 2
Oedema peripheral (General disorders) | 11 | 14 | 11 | 0 | 7
Pain (General disorders) | 6 | 6 | 3 | 0 | 3
Pyrexia (General disorders) | 11 | 9 | 21 | 2 | 8
COVID-19 (Infections and infestations) | 11 | 8 | 7 | 1 | 2
Nasopharyngitis (Infections and infestations) | 8 | 5 | 3 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 5 | 7 | 1 | 1
Urinary tract infection (Infections and infestations) | 8 | 12 | 6 | 1 | 4
Alanine aminotransferase increased (Investigations) | 5 | 9 | 7 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 4 | 2 | 3 | 0 | 4
Blood cholesterol increased (Investigations) | 2 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 3 | 12 | 5 | 0 | 6
Lymphocyte count decreased (Investigations) | 5 | 13 | 5 | 0 | 4
Neutrophil count decreased (Investigations) | 25 | 48 | 31 | 1 | 17
Platelet count decreased (Investigations) | 25 | 43 | 13 | 1 | 15
Weight decreased (Investigations) | 5 | 16 | 10 | 0 | 3
Weight increased (Investigations) | 3 | 5 | 2 | 0 | 4
White blood cell count decreased (Investigations) | 16 | 20 | 21 | 1 | 11
Decreased appetite (Metabolism and nutrition disorders) | 35 | 68 | 41 | 3 | 27
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 9 | 11 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 3 | 5 | 0 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 9 | 11 | 0 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2 | 5 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 10 | 7 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2 | 5 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 17 | 9 | 0 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 13 | 12 | 0 | 4
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 8 | 6 | 0 | 4
Dizziness (Nervous system disorders) | 12 | 11 | 10 | 0 | 5
Dysgeusia (Nervous system disorders) | 19 | 40 | 26 | 0 | 9
Headache (Nervous system disorders) | 7 | 15 | 15 | 1 | 7
Taste disorder (Nervous system disorders) | 4 | 5 | 2 | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 7 | 19 | 5 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 4 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 20 | 9 | 0 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 6 | 1 | 7
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4 | 19 | 8 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 32 | 67 | 0 | 5
Hypertension (Vascular disorders) | 3 | 12 | 6 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2024-05-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT05218499/Prot_003.pdf
  • Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/99/NCT05218499/SAP_004.pdf